CLINICAL TRIAL: NCT05849974
Title: Large Cohort of 1000 Patients With Severe Myopia
Acronym: MyoCo1000
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Collaborators: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P22-03
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-04

CONDITIONS: Myopia, Severe
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Prospective, longitudinal, multicentric, non-randomized cohort study with constitution of a biological collection.
  This study will include major and minor patients with high myopia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hight Myopa (Experimental): Large Cohort of patients with hight Myopa
  Interventions: Other: Structural and fonctional phynotyping

INTERVENTIONS:
Other: Structural and fonctional phynotyping — The additioan acts in this research are:
  Fonctionnal phenotyping:Retinal sensitivity and fixation stability assessment using microperimetry, assessment of long-term fixation stability Structural Phenotyping: Anterior segment examination with OCT anterior Blood sample collection

SUMMARY:
The prevalence of myopia and severe myopia are increasing and will affect 50% and 10% of the population respectively. Severe myopia exposes an increased risk of glaucoma, cataract, retinal detachment and myopic maculopathy, a source of visual impairment.

To date, no European cohort study has been conducted to estimate the rate of these complications and to study the predictive parameters.

DETAILED DESCRIPTION:
This study allows to describe the evolution of different ophthalmological parameters of a population of strong myopes during their follow-up for 10 years using multimodal imaging techniques of the retina.

Prospective, longitudinal, multicentric, non-randomized cohort study with constitution of a biological collection.

This study will include major and minor patients with high myopia

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 6 years
* Severe myopia in at least one eye, defined as

  * a refractive error ≤ -6.00 diopters OR
  * an axial length ≥ 26.50 mm
* Follow-up performed at at least one of the participating centers
* Express consent to participate in the study
* If age < 18 years: express consent of the person(s) exercising parental authority
* Affiliated or beneficiary of a health insurance

Exclusion Criteria:

* Visual acuity < 5 letters on the ETDRS (equivalent to "finger count" or less) in both eyes
* Disorders of the transparent media in both eyes with opacities that may affect image quality
* Syndromic myopia of genetic origin (Stickler syndrome type 1 and 2, Marfan syndrome, Ehler-Danlos disease type 4, Knobloch syndrome) or inherited retinal dystrophy (X-linked retinitis pigmentosa, congenital stationary night blindness of Schubert-Bornshein type, Bornholm eye disease)
* Patient who does not wish to continue to be followed in one of the participating centers
* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding woman

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2038-05 (Estimated); Study Completion 2038-05 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 10 years
  Using the ETDRS and the near vision scale (decimal scales converted to logMAR)
Refraction measures | 10 years
  Measure will be performed in diopter
Lens opacity | 10 years
  Measure will be performed in pixel units
Intraocular pressure and pachymetry | 10 years
  These measurements are respectively carried out in mmHg and in μm
Retinal sensitivity and fixation stability | 10 years
  Respectively Performed in decibels and by microperimetry
Central visual field deficits | 10 years
  by automatic perimetry in decibels
Axial length | 10 years
  Will be performed in mm
Quantitative data | 10 years
  On optical coherence tomography (OCT) and OCT-Angiography
qualitative data on OCT : | 10 years
  presence of any macular complications:
  * condition of the posterior vitreous
  * presence of inner or outer retinal alteration (fluid, layer disorganization, band interruption...).
Area of Rétinal atrophy | 10 years
  In autofluorescence (in mm²)
Characterization of the type of staphyloma | 10 years
  staphyloma classification
Vitreous status | 10 years
  Liquefaction, stage of posterior vitreous detachment
Excavation of the optic nerve and area | 10 years
  In mm² of peripapillary atrophy on color and autofluorescence images
Anterior segment status | 10 years
  Chamber measurement, corneal curvature (in mm)

SECONDARY OUTCOMES:
Macular ophthalmologic complications | 10 years
  Diffuse atrophy/patch atrophy/macular atrophy
  * Choroidal neovessel
  * Bruch's membrane rupture
  * Bulging macula
  * Papillary dysversion
  * Myopic staphyloma
  * Epiretinal membrane
  * Lamellar hole
  * Myopic foveoschisis
  * Macular hole
Non-macular ophthalmologic complications | 10 years
  * Glaucoma optic Neuropathy
  * Cataract
  * Retinal detachment

CONTACTS AND LOCATIONS:
Overall Officials: Ramin TADAYONI, Pr, Principal Investigator — Hôpital Fondation Adolphe de Rothschild